CLINICAL TRIAL: NCT05337774
Title: Imaging [18F]PI-2620 and [18F]Florbetaben in Military Service Members With Blast Related Mild Traumatic Brain Injury
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: study funding period ended March 2022
Sponsor: Life Molecular Imaging SA (Industry)
Collaborators: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-03690
Record Dates: First submitted 2022-02-09; First posted 2022-04-20 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Mild Traumatic Brain Injury
Keywords: Tau PET; [18F]PI-2620; Florbetaben; TBI; Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion; Brain Injuries, Traumatic | interventions — ((18)F)PI-2620

STUDY DESIGN:
Intervention Model Description: This is an exploratory Phase 1, case-control study. Neuroimaging, neuropsychological tests, medical history reviews, and questionnaires will be collected for all eligible subjects.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Blast-related mTBI group (Experimental): Assessments will include:(i) neuropsychological and neurobehavioral testing, (ii) MRI, with a special emphasis on (iii) PET, using emerging tracers for tauopathy ([18F]PI-2620), and amyloid ([18F]florbetaben).
  Interventions: Drug: [18F]PI-2620
- mTBI not blast-related (control group 1) (Experimental): Assessments will include:(i) neuropsychological and neurobehavioral testing, (ii) MRI, with a special emphasis on (iii) PET, using emerging tracers for tauopathy ([18F]PI-2620), and amyloid ([18F]florbetaben).
  Interventions: Drug: [18F]PI-2620
- no history of TBI (control group 2) (Experimental): Assessments will include:(i) neuropsychological and neurobehavioral testing, (ii) MRI, with a special emphasis on (iii) PET, using emerging tracers for tauopathy ([18F]PI-2620), and amyloid ([18F]florbetaben).
  Interventions: Drug: [18F]PI-2620

INTERVENTIONS:
Drug: [18F]PI-2620 — The participant will be injected with 5 mCi (185 MBq) [18F]PI-2620 via a short line which will be placed in an intravenous line in an antecubital vein. Subjects will be placed in the scanner after injection and dynamic scans will be acquired for 0 to 60 minutes post injection.

SUMMARY:
The main objective of this interdisciplinary study is to develop an understanding of the molecular imaging features of blast-related mild traumatic brain injury (mTBI) in military personnel, while helping to establish assessment tools that may be of use in diagnosis, determining prognosis, and in future therapeutic clinical trials. Additionally, the objective is to evaluate feasibility of [18F]PI-2620 in the assessment TBI.

DETAILED DESCRIPTION:
The main objective of this interdisciplinary study is to develop an understanding of the molecular imaging features of blast-related mild traumatic brain injury (mTBI) in military personnel, while helping to establish assessment tools that may be of use in diagnosis, determining prognosis, and in future therapeutic clinical trials. Additionally, the objective is to evaluate feasibility of [18F]PI-2620 in the assessment TBI. This particular tracer has been shown to be effective in localizing tau deposition. [18F]PI-2620 has not yet received FDA approval for routine clinical use and for the purpose of this study is considered an Investigational New Drug (IND) by the FDA.

ELIGIBILITY:
Inclusion Criteria:

1. Male
2. Right-handed
3. Age 25-54
4. Agree to participate in ALL study procedures
5. English speaking
6. Ambulatory
7. Must be able to identify a study partner who is well acquainted with the participant for at least 2 years, to answer questions either in person or over the telephone about the participants' activities of daily living, and to corroborate behavioral and cognitive problems and history of brain injury
8. History of combat deployment
9. For blast-related mTBI group: must be active duty or DEERS-eligible, currently or formerly enrolled in the 4 week intensive outpatient program at NICoE, have experienced 1 or more blast-related mTBIs during tours of duty and report experiencing changes in mood, behavioral or cognitive problems (blast-related mTBI considered here and confirmed in EMR as: blast exposure from explosive device resulting in mTBI which fits criteria defined by VA DoD mTBI guidelines which include at least one of: at time of injury - LOC 0-30 minutes, AOC up to 24hrs, PTA 0-1 day, GCS 13-15)
10. DEERS-eligible for all participants
11. For control group 1: history of mTBI with no blast-related mTBIs (as confirmed in EMR and/or by the BISQ and QCube) 12. For control group 2: No lifetime history of TBI (as confirmed by the BISQ and/or EMR)

Exclusion Criteria:

1. Had a moderate or severe brain injury that required hospitalization
2. Significant systemic illness or unstable medical conditions including: uncontrolled diabetes mellitus, uncorrected hypothyroidism or hyperthyroidism, or systemic cancer
3. Diagnosis of schizophrenia, psychosis, or other psychological disorder (Note: blast-related mTBI group will not be excluded if they have a stable diagnosis of post-traumatic stress disorder, depression and anxiety resulting from their military experience; disorders existing prior to military service will serve as an exclusion)
4. Current and active alcohol or substance abuse or dependence (DSM V criteria) within the past 6 months
5. Clinically significant laboratory test abnormalities (such as hematology, chemistry, urinalysis, ECG) or significant impairment of liver or renal function
6. Significant cerebrovascular disease (such as TIA, stroke) or cardiovascular disease (such as uncontrolled hypertension, atrial fibrillation)
7. Impairment of visual or auditory acuity sufficient to interfere with completion of study procedures
8. Education level < 10 years
9. The presence of any MRI-incompatible prostheses or ferromagnetic metal, or any other condition that would preclude ability to undergo MRI or PET (such as claustrophobia or obesity, >350 lbs and/or unable to fit in scanners)
10. History of risk factors for torsade de pointes or take drugs known to prolong the QT interval
11. Had 2 or more PET scans in the last year, or other significant exposure to radiation (i.e. radiation therapy)
12. Diagnosis of neurodegenerative or neurological diseases and dementia (other than CTE) such as Alzheimer's disease, Parkinson's disease, vascular dementia, Huntington's disease, Pick's disease, Lewy Body Dementia, frontotemporal dementia, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, or multiple sclerosis

Ages: 25 Years to 54 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Due to limited participant availability women will not be included in the study.
Enrollment: 18 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Tau deposition in the brain as measured with PI-2620 PET | 1 day
  Tau deposition in the brain of military personnel with blast-related mTBI, non-blast mTBI or no history of TBI will be measured with PI-2620 using positron emission tomography.
Amyloid deposition in the brain as measured with Florbetaben PET | 1 day
  Amyloid deposition in the brain of military personnel with blast-related mTBI, non-blast mTBI or no history of TBI will be measured with Florbetaben using positron emission tomography.

SECONDARY OUTCOMES:
Correlation of brain MR imaging with PI-2620 brain PET imaging | 1 day
  Brain MR imaging will be performed and results correlated with PI-2620 brain PET imaging
Neurocognitive deficits present in military personnel with blast-related mTBI as measured with NICoE | up to 4 weeks
  Neuropsychology assessment will be performed with NICoE, an intensive outpatient program. All subjects will undergo a battery of standardized questionnaires and neuropsychological tests that will characterize the cohort across multiple neuropsychological domains.

CONTACTS AND LOCATIONS:
Locations (1):
- Walter Reed National Military Medical Center (WRNMMC), Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-02-08): https://cdn.clinicaltrials.gov/large-docs/74/NCT05337774/ICF_000.pdf